CLINICAL TRIAL: NCT04885166
Title: Preventing Prescription Stimulant Diversion and Medication Misuse Via a Web-Based Simulation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity College (Other)
Collaborators: Texas State University (Other); University of Wyoming (Other)
Responsible Party: Principal Investigator, Laura Holt, Associate Professor of Psychology, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R34DA048345-01A1 (NIH)
Record Dates: First submitted 2021-05-04; First posted 2021-05-13 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Prescription Drug Abuse (Not Dependent); Intentional Misuse
Keywords: diversion
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Web-based simulation intervention (Experimental): Participants in this condition will receive psychoeducation about stimulant medication diversion, stimulant medication misuse, and will practice navigating and resisting requests for their medication with a virtual human.
  Interventions: Behavioral: Web-based simulation active intervention
- Placebo condition (Placebo Comparator): Participants in this condition will learn about psychological conditions that affect college students most often (e.g., depression), causes of those conditions, and pharmacological/behavioral treatments for those conditions.
  Interventions: Other: Web-based placebo presentation

INTERVENTIONS:
Other: Web-based placebo presentation — This presentation will discuss the prevalence of psychological disorders in college students, their etiologies, psychiatric medications, and students' personal experiences navigating college with a diagnosis of an anxiety and learning disorder, respectively. Attention-deficit/hyperactivity disorder and stimulant medications will be addressed, but diversion and medication misuse will not be discussed.
  Arms: Placebo condition
Behavioral: Web-based simulation active intervention — This intervention engages students in interactive discussions with virtual humans to (a) learn about the actual prevalence of NMUPS and diversion and their related risks, (b) practice using refusal strategies when approached for their medication in high-risk situations, and (c) understand how to effectively communicate with prescribers and avoid medication misuse.
  Arms: Web-based simulation intervention

SUMMARY:
Half or nearly half of college students with prescriptions divert their stimulant medication, and a similarly high percentage misuse their medication or use someone else's prescription. Diversion may lead students to go without needed medication to mitigate their symptoms, increasing their risk for unintentional injuries and substance use. Further, diversion perpetuates the non-medical use of prescription stimulants (NMUPS), which has become increasingly common among college students. Diversion also perpetuates medical misuse of stimulants among students with prescriptions, which is associated with poorer attention-deficit/hyperactivity disorder (AD/HD) symptom management and may increase the risk for addictive disorders. There are no evidence-based interventions targeting diversion of stimulants in college students. Being approached for one's medication is a key risk factor for diversion, as is medication non-adherence and believing NMUPS and diversion are more prevalent than they are. Accordingly, in this multi-site study, the investigators will conduct a randomized, controlled trial of 300 college-attending adults with current stimulant prescriptions to examine the preliminary efficacy and feasibility of a single-session, computer-based simulation intervention (with two booster sessions) to prevent prescription stimulant diversion and medication misuse and compare it to a placebo condition. The intervention, which is grounded in social learning theory and the theory of planned behavior uniquely engages students in interactive discussions with virtual humans to (a) learn about the actual prevalence of NMUPS and diversion and their related risks, (b) practice using refusal strategies when approached for their medication in high-risk situations, and (c) understand how to effectively communicate with prescribers and avoid medication misuse. The primary aims are to determine if the intervention reduces diversion, intentions to divert, and medication misuse, and to assess user satisfaction with the intervention. The secondary aims are to examine change in potential mechanisms of action targeted in the intervention, such as self-efficacy to resist diversion, knowledge about diversion and NMUPS, use of behavioral strategies to resist requests for one's medication, and prescriber communication. If effective, the intervention could be readily and widely disseminated to college counseling centers, psychiatrists, pediatricians, and other prescribers.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate or graduate student at Trinity College (CT); University of Wyoming; Texas State University.
* Will be enrolled at Trinity College (CT); University of Wyoming; Texas State University 6-months from their baseline study session.
* Have a recent (within the past 3 months) prescription for a stimulant medication
* Between the ages of 17 and 25.

Exclusion Criteria:

* None.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 249 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Change in frequency of prescription stimulant diversion | baseline, 3-months, 6-months
  participants will note how many times they have engaged in diversion (i.e., giving away, selling, or trading one's prescribed medication)
Change in intention to divert prescription stimulant medication | baseline, 3-months, 6-months
  How likely is it that you will give away, sell, or trade your stimulant medication in the next three months?
Change in frequency of prescription stimulant medication misuse | baseline, 3-months, 6-months
  participants will indicate any instances of (a) using alternative routes of administration, (b) taking more than your recommended dose, (c) taking less than your recommended dose, (d) taking someone else's stimulant medication, (e) taking your stimulant with other drugs in order to experience intoxicating effects, or (f) intentionally getting high on your prescribed stimulant medication?
User satisfaction with the simulation/placebo | baseline (immediately after simulation or placebo presentation)
  We will assess the usefulness, information quality, and interface quality of the simulation using the 13-item Post-Study System Usability Questionnaire. A mean score of 1 indicates lowest level of satisfaction, while a mean score of 7 would indicate the highest level of satisfaction.
Usability of the simulation/placebo | baseline (immediately after simulation or placebo presentation)
  Participants will respond to 15 items related to the perceived usefulness, user control, and impact of the simulation/placebo. A mean score of 1 would indicate the lowest level of perceived usability; a mean score of 5 would indicate the highest rating of usability.
1 month booster engagement | 1 month
  We will determine engagement in the online booster session #1 on a 0-5 scale by summing the number of correct answers to the five comprehension questions embedded in the online booster.
2 month booster engagement | 2 months
  We will determine engagement in the online booster session #2 on a 0-5 scale by summing the number of correct answers to the five comprehension questions embedded in the online booster.

SECONDARY OUTCOMES:
Change in self-efficacy to resist prescription stimulant diversion | baseline, 3-months, 6-months
  Participants will rate their confidence to (1) resist giving away their medication, (2) resist selling their medication.
Resistance strategy use | 3- and 6-months
  If, since the last assessment, participants indicate they have been approached for their stimulant medication, they will be asked to describe how they responded (gave/sell/traded medication or not) to each request. In cases where they did not divert their medication, they will be asked to indicate (open-ended response) how they turned down the request.
Change in perceived behavioral norms | baseline, 3-months, 6-months
  Participants will indicate, on a scale from 0-100, what percent of students, on average, engage in (1) diversion and (2) non-medical prescription stimulant misuse.
Change in risk perception | baseline, 3-months
  We will assess perceived legal risks associated with prescription stimulant diversion. We will assess perceived harm from non-medical prescription stimulant use and medical misuse by asking: "How much do people risk harming themselves (physically or in other ways) if they "take stimulants non-medically?" or "use their prescription in a way a prescriber did not intend?
Change in communication with prescriber | baseline, 3-months, 6-months
  Number of times participants communicated with their prescriber regarding their adherence to their prescription and any concerns they have regarding the dose, frequency of administration, and/or side effects in past 90 days.

OTHER OUTCOMES:
Other substance use | baseline, 3-months, 6-months
  Participants will report any occasions of binge drinking, and/or marijuana, cocaine, heroin, methamphetamine, or hallucinogen use, or other prescription drug misuse in the previous 90 days.
Conduct problems | baseline
  Participants will report on the frequency with which they engaged in 11 problem behaviors before age 18
Change in Attention-Deficit/Hyperactivity Disorder-related impairment | baseline, 6-months
  Participants will report on the extent to which they have experienced problems in social, academic, familial, and vocational circumstances. A positive mean change score will indicate that participants experience an increasing level of impairment over the study period, while a negative mean change score will indicate improvement in impairment.
Accidental injuries | 6-months
  Participants will note whether they experienced any accidental injuries in the prior 6 months (e.g., car accidents, burns, etc.).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Trinity College, Hartford, Connecticut
  - Texas State University, San Marcos, Texas
  - University of Wyoming, Laramie, Wyoming

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holt LJ, Looby A, Feinn R, Schepis TS. Preventing Prescription Stimulant Diversion and Misuse via a Web-Based Intervention: A Randomized Controlled Trial. J Atten Disord. 2026 Feb;30(2):265-280. doi: 10.1177/10870547251405545. Epub 2025 Dec 30. PMID 41467299
- [Derived] Holt LJ, Looby A, Schepis TS, Feinn R. Preventing prescription stimulant diversion and misuse through brief intervention: Moderators and secondary outcomes from a randomized controlled trial. Exp Clin Psychopharmacol. 2026 Feb;34(1):61-67. doi: 10.1037/pha0000808. Epub 2025 Nov 10. PMID 41213561